CLINICAL TRIAL: NCT06424132
Title: Identification of Thermogenic Silencing Regulatory Factors as Biomarkers of Metabolic Health in Humans
Brief Title: Thermogenic Silencer Regulatory Factors in Humans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rockefeller University (Other)
Collaborators: Cornell University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PCO1051
Record Dates: First submitted 2024-05-10; First posted 2024-05-21 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Obesity; Metabolic Disease; Cold Exposure
MeSH Terms: conditions — Obesity; Metabolic Diseases | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Intervention Model Description: Participants in from the three different study groups (lean, obese, and obese with type 2 diabetes) will receive the same intervention: cold environmental exposure followed by a rewarming period
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Obese group (Experimental): Body Mass Index (BMI) is > 30, Hemoglobin A1c (HgA1c) <5.7%
  Interventions: Other: Cold Vest Exposure Period; Other: Rewarming Exposure Period; Other: Fasting
- Obese group with Type II diabetes (Experimental): Body Mass Index (BMI) is > 30, Hemoglobin A1c (HgA1c) is >6.5%
  Interventions: Other: Cold Vest Exposure Period; Other: Rewarming Exposure Period; Other: Fasting
- Lean group (Experimental): Body Mass Index (BMI) is between 18.5 and 24.9. Hemoglobin A1c (HgA1c) <5.7%
  Interventions: Other: Cold Vest Exposure Period; Other: Rewarming Exposure Period; Other: Fasting

INTERVENTIONS:
Other: Cold Vest Exposure Period — A cold vest will be placed on the participant which consists of a water-perfused wearable vest, size S-M or M-L with adjustable straps attached to a small 'cooler' reservoir to circulate cold water between the vest and the cooler (Polar Products, Stow, OH- Product link: www.polarproducts.com/polarshop/pc/CoolOR-13-Quart-System-with-Arctic-Chiller-p24757.htm) This product is safe and recommended by experimental guidelines for human BAT studies. Participants will be cold exposed for a period of 3 hours resting in a reclined position engaged in reading and/or digital entertainment of their choice.
Other: Rewarming Exposure Period — Following cold exposure, the cold vests will be removed, and participants will be offered a warm blanket to ease the transition from cold back to warm temperatures. Participants will then be moved to an adjacent warm room maintained at 30 degrees celsius and asked to return to the resting position of their choice. Participants will then engage in reading and/or digital entertainment for a 3-hour warm exposure period.
Other: Fasting — Participants will be requested to refrain from food and caloric drinks for 12 hours (starting at 8pm) prior to the study visit. Blood will then be drawn the following morning (between 8 and 9am) 30mins later following a breakfast meal (9:30am- 10am). Participants will be housed in a room with ambient temperature at 25 degrees celsius between the two blood draws.

SUMMARY:
A promising approach to correct the metabolic dysfunction associated with obesity is to activate brown fat non-shivering thermogenesis (NST). A critical limitation with NST as a therapeutic option, however, is that this beneficial process is silenced under human physiological temperature conditions and the mechanisms of how this occurs is unknown. This study will be the first to identify human NST silencing factors that may be targeted for the treatment of obesity and metabolic disorders.

DETAILED DESCRIPTION:
Obesity and associated metabolic diseases such as type 2 diabetes continue to be one of the leading causes of death worldwide, demanding additional research into novel treatments beyond our current options. One promising experimental approach to overcome the metabolic dysfunctions associated with obesity, such as insulin resistance and glucose imbalance, is to activate brown fat non-shivering thermogenesis (NST). Activated human brown adipose tissue (BAT) increases energy expenditure at a molecular level and is associated with both improved insulin tolerance and glucose homeostasis. A critical limitation with human brown fat as a therapeutic option, however, is that its beneficial metabolic potential is restricted in a silenced state under physiological temperature conditions for most of human life. The regulatory factors that govern this silencing process are completely unknown. While many groups continue to seek novel mechanisms to activate brown fat, this study presents a unique approach, aiming to decipher the mechanisms that govern human brown fat silencing. The study hypothesizes that if the regulatory factors that silence brown fat NST can be defined, then these factors can be targeted for ablation to eliminate the "off switch", thereby keeping brown fat in a constitutively active state. Identification of human NST silencing factors will be critical to unlocking the metabolic benefits of human brown fat and would represent promising treatment opportunities for type 2 diabetes and other obesity-related disorders. Understanding these relationships will allow for precision treatment opportunities for type 2 diabetes in the future.

The overall goal of this study is to unlock the metabolic benefits of human brown fat by defining the regulatory mechanisms that keep BAT in a silenced state. The study will generate the first human secretome (list of secreted proteins in blood) and transcriptome (list of gene transcripts in adipose tissue) compendium from human plasma and subcutaneous adipose tissue respectively which will be composed of target proteins, metabolites, and genes that are differentially expressed in response to NST silencing conditions. Top candidates from the profiling will then be functionally validated in human adipocytes for their role in NST silencing. The study will be an important resource for the field and will identify novel candidates that may harbor regulatory potential to govern the NST silencing process in humans. These factors can then be targeted to promote the constitutive activation of NST in order to overcome the metabolic dysfunction associated with obesity and metabolic disease. Given the invasive nature of direct human brown fat sampling, the study will instead interrogate circulating factors in human plasma as a proxy for metabolic health. In addition, the study will also obtain subcutaneous adipose tissue for RNA profiling to identify genes that are upregulated under NST-silenced conditions compared to cold exposure.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 years old and 35
2. Lean group: BMI is between 18.5 and 24.9. HgA1c <5.7%
3. Obese group: BMI is >30, HgA1c <5.7%
4. Obese group with Type II diabetes: BMI is >30, HgA1c is >6.5% If on oral medication for diabetes management, HgA1c may be < 6.5% The following medications are also acceptable: statins, aspirin, angiotensin-converting enzyme inhibitors (ACEi), and angiotensin receptor blockers (ARB).

Exclusion Criteria:

1. Diabetes type I (self-report)
2. Diagnosis of thyroid disease (including goiter, hyperthyroidism, hypothyroidism, thyroiditis)(self-report)
3. Diagnosis with cancer including skin cancer (self-report)
4. Diagnosis or evidence of Raynaud's Syndrome or systemic sclerosis (self-report)
5. A recent diagnosis of Coronavirus Disease 2019 (COVID-19) (last 2 weeks) or hospitalized at the time of diagnosis with COVID-19
6. Any vaccine administration within two weeks preceding the study procedure
7. Currently pregnant
8. Currently taking any prescribed medication other than oral contraceptives. Treatments for weight loss or any other supplements that may alter weight or metabolism are not acceptable. Vitamins are acceptable.
9. Has consumed nicotine (smoking, inhaling, ingesting) within the last 6 months
10. Has used illicit drugs within the last 6 months (marijuana users are eligible unless consumed in the last 30 days).
11. Any medical, psychological, or social condition that, in opinion of principle investigators, would jeopardize the health or well-being of the participant during the study procedure or the integrity of the data
12. Diabetes Type II that is managed by insulin.
13. Steroid use in the last 30 days to the exclusions

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Identification of adipose tissue transcriptome | Before and after 3-hour rewarming period.
  RNA sequencing to measure and identify a list of gene transcripts that are differentially expressed before and after re-warming. A true change is defined as 1.5 fold increase or decrease in gene expression.
Identification of cold and warm-regulated proteome. | Before and after 3 hour cold exposure period and before and after 3 hour rewarming period.
  Proteins will be captured from blood and analyzed via mass spectrometry which generates a list of proteins for each sample. The investigators will compare the mean fold change (true change is greater than 1.5 fold) in protein abundance at the specified study time points.
Identification of cold and warm-regulated metabolome. | Time frame will be before and after 3 hour cold exposure period as well as before and after 3 hour rewarming period.
  Metabolites will be captured from blood and analyzed via mass spectrometry which generates a list of metabolites for each sample. The investigators will compare the mean fold change (true change is greater than 1.5 fold) in metabolite abundance at the specified study time points.

SECONDARY OUTCOMES:
Nutritional assessments of individuals correlated to expression patterns of human silencer regulatory factors. | Baseline
  Diet History Questionnaire III (DHQ III) to assess food consumption patterns as it relates to the Dietary Guidelines for Americans.
Body Mass Index (BMI) correlated to expression patterns of human silencer regulatory factors. | Baseline
  BMI is calculated by weight and height measured by anthropometric assessments, using the formula weight in kilograms divided by height in meters squared (kilograms/meter^2).
Fat mass body composition (%) measured by Bod Pod correlated to expression patterns of human silencer regulatory factors. | Baseline
  Bod Pod uses Air Displacement Plethysmography (ADP) to determine body composition, the ratio of fat mass to lean mass. The investigators will measure fat mass composition in units of percentage (%).
Lean Mass body composition (%) measured by Bod Pod correlated to expression patterns of human silencer regulatory factors. | Baseline
  Bod Pod uses Air Displacement Plethysmography (ADP) to determine body composition, the ratio of fat mass to lean mass. The investigators will measure lean mass composition in units of percentage (%).

CONTACTS AND LOCATIONS:
Overall Officials: Joeva Barrow, Ph.D., R.D., Principal Investigator — The Rockefeller University and Cornell University; Paul Cohen, Ph.D., M.D., Principal Investigator — The Rockefeller University
Locations (1):
- Rockefeller University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-15): https://cdn.clinicaltrials.gov/large-docs/32/NCT06424132/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-15): https://cdn.clinicaltrials.gov/large-docs/32/NCT06424132/ICF_001.pdf